CLINICAL TRIAL: NCT06845566
Title: Formulation of a Novel Compensation Based Intervention to Improve Activities of Daily Living: A Randomized Controlled Pilot Study
Brief Title: Formulation of Compensation Based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Kaya Ozturk, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HÜ-OT-LKO-03
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: activities of daily living; stroke; compensatory; problem solving; participation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Two groups with an intervention group and a control group
Who Masked: Outcomes Assessor
Masking Description: The therapist who conducted the assessment tests was unaware of the participants' group assignments (interventon or control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (intervention group) (Active Comparator): The intervention group received both compensation-bocused problem-solving therapy and standard rehabilitation services. Standard Rehabilitation:The program allows individuals to utilize the physiotherapy and occupational therapy units on a weekly basis, with access available on weekdays. Compensation Based Problem Solving Therapy (CFPS) is an approach based on the occupational adaptation model. It entails the implementation of compensatory strategies with the objective of enhancing the performance of both extremities in activities of daily living.
  Interventions: Behavioral: Compensation Based Problem Solving Therapy; Behavioral: standard rehabilitation
- Plasebo (control group) (Active Comparator): The control group received standard rehabilitation services. Standard Rehabilitation:The program allows individuals to utilize the physiotherapy and occupational therapy units on a weekly basis, with access available on weekdays
  Interventions: Behavioral: standard rehabilitation

INTERVENTIONS:
Behavioral: Compensation Based Problem Solving Therapy — Compensation-Based Problem Solving Therapy (CB-PST) is a therapeutic approach based on the occupational adaptation model. It entails the implementation of compensatory strategies with the objective of enhancing the performance of both extremities in daily life activities. The therapy encompasses the implementation of problem-solving training. The occupational problem is defined. The development of compensation-focused strategies is based on the "personal factors" and "occupational environment" identified as relevant to the problematic occupation, as determined according to the principles of the occupational adaptation model. Once a compensatory strategy has been selected, the next step is to apply it and evaluate its efficacy, with the expectation that an "adaptive response" will be observed, and that the resulting adaptation will be reflected in improved occupational performance, as guided by the occupational adaptation model.
  Arms: Aspirin (intervention group)
Behavioral: standard rehabilitation — The standard rehabilitation program is provided to all individuals in the inpatient service on an equal basis. The program allows individuals to utilize the physiotherapy and occupational therapy units on a weekly basis, with access available on weekdays. These units are staffed by physiotherapists and occupational therapists. All individuals included in the study received the same service from the same therapists at the same times in a homogeneous manner. All individuals received physiotherapy, electrotherapy, and hydrotherapy as part of this service. In the physiotherapy unit, the first intervention was 25 minutes of electrotherapy for the upper extremity. This was followed by 40 minutes of physiotherapy exercises, conducted with the assistance of a physiotherapist. The final component of the physiotherapy unit programme was 15 minutes of hydrotherapy. In the occupational therapy unit, a standard 40-minute occupational therapy was completed

SUMMARY:
The primary aim of this study was to pilot CBPST as a novel intervention method. By applying it to a pilot group, the research sought to contribute to the existing literature by offering a compensation-based rehabilitation approach

DETAILED DESCRIPTION:
The study was designed as prospective and a randomized controlled pilot study. A simple randomization method was employed to randomly assign individuals to two groups (intervention and control groups). A simple randomization method was employed, whereby the intervention and control group papers were selected from a closed envelope. Following the initial evaluation of each participant, one of the papers bearing the designation "intervention" or "control" was selected at random. This decision determined whether the individual would be included in the intervention or control group. The study was conducted in the occupational therapy department of the physical therapy and rehabilitation clinic of Etlik City Hospital. The study was approved by the Ethics Committee of Etlik City Hospital and was assigned the code AEŞH-EK-2025-025. Following approval from the ethics committee, the Compensation-Based Problem Solving Training (CBPST) was developed. The training program was developed in accordance with the tenets of the Occupational Adaptation Model. All subsequent steps were conducted in accordance with the aforementioned model. The adaptive response, as outlined in the model, encompasses the occupational adaptation that is anticipated to occur at the conclusion of the training program. The therapy was then trialled with a pilot group of five individuals, with the aim of refining the content. Subsequently, the final iteration of the training program was established. All individuals included in the study signed a consent form indicating their willingness to participate. This was completed at the outset of the study. All individuals were provided with a standard rehabilitation program comprising five days a week (40 minutes) of routine therapy. In addition to this, the intervention group received CBPST in the form of five days a week (20 minutes) sessions. The evaluations completed at the beginning of the training were repeated one month later.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of ischemic stroke due to a middle cerebral lesion,
* age between 18 and 64 years,
* a score of 24 or above on the Standardized Mini-Mental State Examination --
* willingness to participate in the study.

Exclusion Criteria:

* Stroke onset between 3 and 12 months prior to the study,
* presence of aphasia (speech impairment)
* diagnosis of another chronic condition that could affect study outcomes

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
The Canadian Occupational Performance Measure (COPM) | 1 month
  It is a scale that includes a semi-structured interview. Activities that individuals have problems with or want to do in self-care, work and productive activities, and leisure activities are determined and given importance points. Then, the most important activities are ranked, and performance and satisfaction points are requested.These scores are made between 0 and 10. The final score is determined by adding the maximum of five activity, performance, and satisfaction scores. The validity and reliability of the scale have been established in the Turkish context.

SECONDARY OUTCOMES:
Functional Independence Scale (FIM) | 1 month
  It is a particularly noteworthy instrument. The FIM was developed to measure independence in daily living activities. The FIM comprises two sub-domains: motor and cognitive status, each with 18 items. The motor sub-domain encompasses 13 items, including feeding, bathing, and transferring, while the cognitive sub-domain comprises 5 items such as understanding, expressing, and social participation. Each item is scored on a scale ranging from 1 to 7, with higher scores indicating greater independence. A standardized guideline exists to facilitate the scoring process. Scores obtained are indicative of functionality levels. A Turkish validity and reliability study has been conducted.

OTHER OUTCOMES:
Lawton-Brody Instrumental Activities of Daily Living (Lawton-Brody IADL) | 1 month
  scale is a measurement tool designed to assess the performance of activities that are essential to daily living. The instrument was developed to measure instrumental activities of daily living. This instrument is frequently utilized in clinical settings and scientific publications. The scale comprises eight items, including telephone use, transportation, housework, shopping, financial management, and medication adherence. Each item is scored on a scale of 0 to 1. Higher scores indicate higher functionality. A Turkish validity and reliability study has been conducted.
Frenchay Activities Index (FAI): | 1 month
  It is another scale that has been utilized in clinical and literary studies. It comprises eight items, including telephone use, transportation, housework, shopping, financial management, and medication adherence. Each item is scored on a scale of 0 to 1, with higher scores indicating better functionality. The FAI is a scale that examines how often one participates in activities of daily living. The index is comprised of 15 items in total. Each item is scored on a scale ranging from 0 to 3, with higher scores indicating greater frequency of participation. Higher scores indicate higher frequencies of engagement in activities. A validity and reliability study has been conducted in Turkish.

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Traning and Research Hospital, Mardin, Artuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No